CLINICAL TRIAL: NCT01051570
Title: Phase II Trial of Carboplatin and Everolimus (RAD001) in Metastatic Castrate Resistant Prostate Cancer (CRPC) Pretreated With Docetaxel Chemotherapy.
Brief Title: Carboplatin, Everolimus, and Prednisone in Treating Patients With Metastatic Prostate Cancer That Progressed After Docetaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000663630; P30CA022453 (NIH); WSU-2009-087; NOVARTIS-WSU-2009-087
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: hormone-resistant prostate cancer; recurrent prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Everolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin, RAD 001 & Prednisone (Experimental): Carboplatin: AUC=4 by Calvert's formula (max dose 600 mg)*IV over 30-60 min, Day 1 of a 21 day cycle
  RAD 001: 5 mg Orally daily, starting from Day 2 continuously
  Prednisone 5 mg Orally twice daily, continuously
  Interventions: Drug: carboplatin; Drug: RAD 001; Drug: prednisone; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: carboplatin — AUC = 5 by Calvert's formula, day 1 of each 21 day cycle
  Other Names: Paraplatin®
Drug: RAD 001 — 5 mg orally starting on Day 2 then continuous
  Other Names: Afinitor®; Zortress; Everolimus
Drug: prednisone — 5 mg orally twice a day starting on Day 1 then continuous
  Other Names: Deltasone; Liquid Pred; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS
Other: laboratory biomarker analysis — Samples will be collected from archival tissue.
Other: pharmacological study — Samples will be collected Cycle 1, day 1, 2 & 8 and Cycle 2, Day 1 & 2

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving carboplatin together with everolimus and prednisone may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin together with everolimus and prednisone works in treating patients with metastatic prostate cancer that progressed after docetaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the time to progression (TTP) achieved with carboplatin and everolimus in patients with castrate resistant metastatic prostate cancer that progressed after docetaxel-based chemotherapy.

Secondary

* To evaluate the safety of this regimen.
* To assess the PSA response rate in patients treated with this regimen.
* To evaluate the overall survival (OS) outcome in these patients.
* To investigate the association of TTP and PSA response rate with correlative markers, such as phospho mTOR, pAKT, and p70S6.
* To evaluate the pharmacokinetics of this regimen.
* To explore the association of TTP, OS, and circulating tumor tumor cell count.

OUTLINE: Patients receive carboplatin IV over 30-60 minutes on day 1, oral prednisone twice daily on days on days 1-21, and oral everolimus once daily on days 2-21 of course 1 and on days 1-21 of subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples are collected periodically for pharmacodynamic, pharmacokinetic, and biomarker analysis.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the prostate
* Objective disease progression or rising PSA despite androgen deprivation therapy and antiandrogen withdrawal (when applicable)
* Progressed after ≥ 1 prior docetaxel-based chemotherapy regimen for metastatic disease

  * Patients with measurable disease* must have either rising PSA, increase in size of the lesion(s), or both

    * Patients with rising PSA as the only evidence of disease progression must demonstrate a rising trend with 2 successive elevations ≥ 1 week apart
  * Patients with no measurable disease must have a PSA ≥ 5 ng/mL or new areas of bony metastases on bone scan NOTE: *There is no minimum PSA requirement for patients with measurable disease
* Documented to be castrate with a testosterone level of ≤ 0.5 ng/mL

  * Leuteinizing hormone-releasing hormone agonist therapy must be continued, if required to maintain castrate levels of testosterone
* No uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Calculated creatinine clearance ≥ 50 mL/min OR serum creatinine ≤ 2 mg/dL
* AST and/or ALT ≤ 2.5 times ULN if alkaline phosphatase normal OR alkaline phosphatase ≤ 4 times ULN if AST and/or ALT normal (for patients without documented bone metastases or for patients with liver metastases)
* AST and/or ALT < 2.5 times ULN, without regard to alkaline phosphatase levels (for patients with documented bone metastases)
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 times ULN (in the case that one or both of these thresholds are exceeded, the patient is eligible only after initiation of appropriate lipid-lowering medication)
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* Willing and able to comply with this study
* Able to ingest oral medication
* No other malignancies except non-melanoma skin cancer or any other adequately treated cancer in complete remission for ≥ 2 years
* No significant traumatic injury within the past 4 weeks
* No active (acute or chronic) or uncontrolled severe infections
* No severe and/or uncontrolled medical conditions or other conditions that could affect study participation, including the following:

  * NYHA class III-IV symptomatic congestive heart failure
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within the past 6 months, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Severely impaired lung function as defined by spirometry and DLCO that is 50% of the normal predicted value and/or oxygen saturation that is ≤ 88% at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 times ULN
  * Liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
  * Known history of HIV seropositivity, hepatitis B or C
  * Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
  * Active, bleeding diathesis
* No known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to their excipients
* No history of noncompliance to medical regimens
* No uncontrolled diabetes mellitus

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 1 prior docetaxel based regimen for metastatic disease

  * Docetaxel based combination therapy or docetaxel alone considered as 1 regimen
* No more than 2 prior chemotherapy regimens for metastatic disease
* No prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus)
* At least 6 weeks since prior bicalutamide or nilutamide
* At least 4 weeks since prior flutamide
* More than 4 weeks since prior and no other concurrent investigational drugs
* More than 4 weeks since prior and no other concurrent anticancer therapies (including chemotherapy, radiotherapy, or antibody-based therapy)
* More than 4 weeks since prior and no concurrent major surgery (defined as requiring general anesthesia) and recovered
* More than 1 week since prior and no concurrent immunization with attenuated live vaccines
* No concurrent chronic, systemic treatment with corticosteroids or other immunosuppressive agents

  * Topical or inhaled corticosteroids are allowed
* No concurrent prophylactic growth factors
* Concurrent bisphosphonate therapy allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - Northshore University Health System, Evanston, Illinois
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey

REFERENCES:
- [Derived] Vaishampayan U, Shevrin D, Stein M, Heilbrun L, Land S, Stark K, Li J, Dickow B, Heath E, Smith D, Fontana J. Phase II Trial of Carboplatin, Everolimus, and Prednisone in Metastatic Castration-resistant Prostate Cancer Pretreated With Docetaxel Chemotherapy: A Prostate Cancer Clinical Trial Consortium Study. Urology. 2015 Dec;86(6):1206-11. doi: 10.1016/j.urology.2015.08.008. Epub 2015 Sep 12. PMID 26375845
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin, RAD 001 & Prednisone: Carboplatin: AUC=4 by Calvert's formula (max dose 600 mg)*IV over 30-60 min, Day 1 of a 21 day cycle
  RAD 001: 5 mg Orally daily, starting from Day 2 continuously
  Prednisone 5 mg Orally twice daily, continuously
  carboplatin: AUC = 5 by Calvert's formula, day 1 of each 21 day cycle
  RAD 001: 5 mg orally starting on Day 2 then continuous
  prednisone: 5 mg orally twice a day starting on Day 1 then continuous
  laboratory biomarker analysis: Samples will be collected from archival tissue.
  pharmacological study: Samples will be collected Cycle 1, day 1, 2 & 8 and Cycle 2, Day 1 & 2
Period: Overall Study
Arm/Group | Carboplatin, RAD 001 & Prednisone
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 69 [54 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Progression defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 63 days while on treatment, then up 90 days thereafter. From date of registration to date of progressive disease.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 26
months | 2.5 [1.8 to 4.3]

2. Secondary Outcome: Number of Participants With Toxicity as Measured by NCI CTCAE v3.0 Criteria
Description: Number of Participants with Grade 3/4 Toxicity as measured by NCI CTCAE v3.0 criteria
Time Frame: Day 1 of each cycle (every 21 days), through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 26
Participants
  Anemia | 10
  Thrombocytopenia | 9
  Lymphopenia | 6
  Leukopenia | 4
  Infection without neutropenia | 4
  Hypophosphatemia | 4
  Neutropenia | 3
  Dehydration | 3
  Hyperglycemia | 3
  Hyponatremia | 3
  Pulmonary embolism | 2
  Fatigue | 2
  Hypercholesterolemia | 1
  Rash | 1
  AST | 1
  Hypomagnesemia | 1
  Hypokalemia | 1

3. Secondary Outcome: PSA Response Rate
Description: PSA response rate with response defined as => a 30% reduction in PSA
Time Frame: Day 1 of each cycle (every 21 days), through study completion, an average of 6 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 26
percentage of participants | 15 [7 to 30]

4. Secondary Outcome: Association of PSA Response Rate With Correlative Markers (Phospho mTOR, pAKT, and p70S6)
Description: PSA response defined as a decrease of 30% or more will be tabled against mTOR, pAKT, and p70S6 (1+, 2+, 3+ vs ND)
Time Frame: Archival tissue will be collected if available. Optional biopsies pre-treatment and 24 hours after first everolimus and carboplatin dose
Population: There were only 2 responders of the 10 participants who were measured for mTOR, pAKT, and p70S6.
Measure: Number; unit: participants
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 2
participants
  pAKT(ND) vs Responder | 1
  mTOR(ND) vs Responder | 0
  p70S6(ND) vs Responder | 1

5. Secondary Outcome: Pharmacokinetics: Observed Carboplatin AUC Was Estimated Based on the Concentration in the 2.75-h Sample.
Description: Using a limited sampling model (i.e., AUC = 0.52 × C2.75h + 0.92) (Sorensen et al., 1993), observed carboplatin AUC was estimated based on the concentration in the 2.75-h sample.
Time Frame: Samples were collected Cycle 2, Day 1
Population: Limited PK sampling for carboplatin were obtained at 2.75 and 24 h after the end of infusion from 8 patients.
Measure: Mean (Full Range); unit: mg/ml*min
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 8
mg/ml*min | 5.8 [4.1 to 11.0]

6. Secondary Outcome: Overall Survival
Description: Overall Survival as measured by the Kaplan-Meier method
Time Frame: After treatment, participants will be contacted every 3 months up to 4 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Carboplatin, RAD 001 & Prednisone
Number analyzed (Participants) | 26
months | 12.5 [7.7 to 18.7]

ADVERSE EVENTS:
Arm/Group | Carboplatin, RAD 001 & Prednisone
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, RAD 001 & Prednisone (N=26)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Dehydration (Gastrointestinal disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Fatigue (General disorders) | 2 (2)
Thrombosis_PE (Vascular disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
AST (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Inf_wo_neutropenia (Blood and lymphatic system disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, RAD 001 & Prednisone (N=26)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Edema (Blood and lymphatic system disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12)
Proteinuria (Metabolism and nutrition disorders) | 11 (11)
Fatigue (General disorders) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
AST (Blood and lymphatic system disorders) | 7 (7)
Creatinine (Metabolism and nutrition disorders) | 6 (6)
Sensory_Neuropathy (Nervous system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 14 (14)
Hypercholesterolemia (Metabolism and nutrition disorders) | 17 (17)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 12 (12)
Inf_wo_neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Small sample size; Correlates were conducted in <50% of the patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No